CLINICAL TRIAL: NCT05639231
Title: Impact of an INtervention TO Increase MOBility in Older Hospitalized Medical Patients (INTOMOB): a Cluster Randomized Controlled Trial
Brief Title: An INtervention TO Improve MOBility of Older Hospitalized Patients
Acronym: INTOMOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other); Hôpital Fribourgeois (Other); Kantonsspital Baden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-01568
Record Dates: First submitted 2022-11-28; First posted 2022-12-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Hospital Mobility; Mobility Limitation; Life-Space; Functional Status; Hospital-Acquired Condition; Muscle Atrophy or Weakness; Sarcopenia; Iatrogenic Disease
Keywords: Hospital mobility; Life-Space; Functional status; Hospital-Acquired disability; Exercise; Movement; Ambulation
MeSH Terms: conditions — Mobility Limitation; Iatrogenic Disease; Muscular Atrophy; Asthenia; Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: In a first phase, the intervention will be pilot-tested in one ward of each hospital (no comparison group).
  In a second phase, it will be tested in a parallel design (cluster randomized controlled trial).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Complete blinding is difficult due to the nature of the intervention and the design (cluster randomization).
  To preserve blinding as much as possible, several strategies have been set.
  At the cluster level (healthcare professional intervention): Since rotation across wards happens at the physician level, but is rare at the level of the nursing staff, the healthcare professional intervention targets mostly nurses. The healthcare professionals will be informed to avoid speaking about the intervention with colleagues of other wards.
  At the patient level, differential information for candidates for the intervention or for the control group (the randomization group is known when first approaching candidates for participation because of the cluster design) will be provided. Candidates for the control group will receive only partial information without explaining the intervention. They will be informed orally at the end of the study about all aspects of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTOMOB intervention (Experimental): The intervention will be multilevel, targeting the patients, healthcare professionals (HCPs) and environment, as described under "Intervention description".
  Interventions: Behavioral: INTOMOB intervention
- Control (No Intervention): Control procedure in the randomized trial:
  * Patients will receive standard of care, including physiotherapy if prescribed by the hospital physician and usual mobility recommendations and support by the HCPs.
  * HCPs will neither complete the e-learning, nor receive the checklist and the oral presentation.
  * The environment will not be modified in regards to mobility. Already existing information on this topic (e.g., small posters hanging in patient rooms) will not be removed, since it corresponds to current standard of care in some hospitals.
  In the pilot study, there will be no control procedure, since the objective is to assess experience and feasibility of the intervention, not its effects.

INTERVENTIONS:
Behavioral: INTOMOB intervention — The intervention will be multilevel, targeting the patients, healthcare professionals (HCPs) and environment:
  PATIENTS:
  * Information booklet on the importance/benefits of mobility, consequences of low mobility, how to be more active (with concrete information).
  * Customizable diary to document mobility goals, results, difficulties and needs.
  * Exercise booklet with explanations & pictures of mobility exercises (supine, sitting, standing).
  * iPad 10.2'' with videos of the exercises.
  HCPs (physicians & nursing staff):
  * E-learning on the consequences of low mobility, barriers/facilitators to hospital mobility; recommendations, documentation, communication & interdisciplinary collaboration regarding mobility; implementation.
  * Oral presentation on the intervention.
  * Checklist to remind HCPs to address mobility.
  ENVIRONMENT:
  * Posters in the wards about mobility and other topics of interest to older adults.
  * Walking itineraries in the wards.
  Arms: INTOMOB intervention

SUMMARY:
Low mobility during an acute care hospitalization is very frequent, particularly among older patients, and associated with adverse outcomes, such as persistent functional decline, institutionalization and death. However, increasing hospital mobility remains challenging because of the multiple existing barriers.

The goal of this clinical trial is to test the effect of a multilevel intervention to increase hospital mobility, which addresses modifiable barriers and facilitators and does not require unavailable additional resources.

This study aims to answer whether this intervention can improve mobility and patient-relevant outcomes such as life-space mobility and functional status.

The multilevel intervention will target:

1. The patients, who will receive an information booklet, a customizable diary, an exercise booklet and an iPad with access to the videos of the exercise booklet.
2. The healthcare professionals (nursing staff and physicians) who will complete an e-learning, receive an oral presentation on the intervention, and receive a "mobility checklist" that reminds them of what they should assess daily regarding mobility.
3. The hospital environment, where posters will be hung in the wards, including walking itineraries, on topics of interest to older adults.

In a first phase, the intervention will be pilot-tested in one ward of each hospital. The intervention will then be adapted based on patient and healthcare professional feedback.

In a second phase, the intervention will be tested in a cluster randomized controlled trial, and compared to standard of care.

ELIGIBILITY:
Inclusion criteria:

* Admission to a general internal medicine (GIM) ward of a participating hospital
* Age ≥60 years
* Being ambulatory during the 2 weeks before admission (self-report)
* Living in the community (not in a nursing home or another institution) for at least the last 30 days prior to admission
* Ability to understand French or German
* Planned length of stay at least 3 days after enrollment
* For the pilot-study only: Possibility to start the study within 48 hours after admission to the GIM ward

Exclusion criteria:

* Medical contraindication to walk (e.g., wound not allowing loading weight)
* Wheelchair-bound
* End-of-life
* Severe psychiatric disorder (severe depression, schizophrenia, psychosis)
* Delirium (according to the Confusion Assessment Method [CAM])

Additional exclusion criterion for the pilot-study only:

- Dementia (defined as Mini-Cog <3)

Additional exclusion criteria for the RCT only:

* Cognitive impairment making impossible to use study material (=implement the intervention) and to understand and sign informed consent, based on clinical judgement, except if a proxy can be actively involved in the study and provides consent
* Severe visual impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Life-space level | Day 30 (+/-5) after enrollment
  Measured by the University of Alabama at Birmingham Study of Aging Life-Space Assessment (range 0-120, with maximum being a higher score = better outcome). For patients institutionalized, assessment through the Life-Space Assessment in Institutionalized Settings. Both scales can be merged since the scoring is similar. Assessment by telephone interview of the participant/relatives.

SECONDARY OUTCOMES:
Life-space level | Day 180 (+/-5) after enrollment
  Measured by the University of Alabama at Birmingham Study of Aging Life-Space Assessment (or Life-Space Assessment in Institutionalized Settings for institutionalized patients) by telephone interview of the participant/relatives
Activities of Daily Living | Day 30 (+/-5) after enrollment
  Measured by the Barthel Index by telephone interview of the participant/relatives
Activities of Daily Living | Day 180 (+/-5) after enrollment
  Measured by the Barthel Index by telephone interview of the participant/relatives
Instrumental Activities of Daily Living | Day 30 (+/-5) after enrollment
  Measured by the Lawton Index by telephone interview of the participant/relatives
Instrumental Activities of Daily Living | Day 180 (+/-5) after enrollment
  Measured by the Lawton Index by telephone interview of the participant/relatives
Quality of life (EQ-5D) | Day 30 (+/-5) after enrollment
  Measured by the European Quality of Life-5 Dimensions (EQ-5D) questionnaire by telephone interview of the participant/relatives
Quality of life (EQ-5D) | Day 180 (+/-5) after enrollment
  Measured by the European Quality of Life-5 Dimensions (EQ-5D) questionnaire by telephone interview of the participant/relatives
Depression | Day 30 (+/-5) after enrollment
  Measured by the Patient Health Questionnaire (PHQ)-2 by telephone interview of the participant/relatives
Depression | Day 180 (+/-5) after enrollment
  Measured by the Patient Health Questionnaire (PHQ)-2 by telephone interview of the participant/relatives
Pressure ulcer | Discharge (-1 to +2 days after discharge)
  Evaluated according to the NPUAP/EPUAP classification, based on nurse report and electronic health record
Delirium during hospitalization (hospitalization duration expected to be 3 to 20 days on average) | Discharge (-1 to +2 days after discharge)
  Measured by the Confusion Assessment Method
Mobility at discharge | Discharge (maximum 1 day before)
  Measured by the de Morton Mobility Index (DEMMI); assessment conducted by the study team
Lower-limb muscle strength | Discharge (maximum 1 day before)
  Measured by lower-limb manual testing according to the method by Hislop and Montgomery; assessment conducted by the study team
Hand-grip muscle strength | Discharge (maximum 1 day before)
  Measured by JAMAR (for the pilot study) and SAEHAN (for the RCT) hand dynamometer; assessment conducted by the study team
Step count during hospitalization (hospitalization duration expected to be 3 to 20 days on average) | Discharge (hospitalization duration expected to be 3 to 20 days on average)
  Measured by a StepWatch ankle accelerometer or a GENEActiv wrist accelerometer (the choice of the device will be defined after the pilot study during which both accelerometers will be tested)
Level of activity during hospitalization (hospitalization duration expected to be 3 to 20 days on average) | Discharge (hospitalization duration expected to be 3 to 20 days on average)
  Measured by GENEActiv wrist accelerometer (only if this accelerometer is chosen after the pilot study)
Fear of / concerns about falling | Discharge (-1 to +2 days after discharge)
  Measured by the Falls Efficacy Scale - International by telephone interview of the participant/relatives
Fear of / concerns about falling | Day 30 (+/-5) after enrollment
  Measured by the Falls Efficacy Scale - International by telephone interview of the participant/relatives
Fear of / concerns about falling | Day 180 (+/-5) after enrollment
  Measured by the Falls Efficacy Scale - International by telephone interview of the participant/relatives
Fall-risk increasing drugs | Discharge (discharge letter) (hospitalization duration expected to be 3 to 20 days on average)
  Including loop diuretic, beta blocker, cardiac glycoside (digitalis, digoxin), statin, antipsychotic (neuroleptic), tricyclic antidepressant, selective serotonin reuptake inhibitor, other antidepressant, benzodiazepine, opioid, antiepileptic. Assessed through the electronic health record
Fall-risk increasing drugs during hospitalization | Discharge (discharge letter) (hospitalization duration expected to be 3 to 20 days on average)]
  Including loop diuretic, beta blocker, cardiac glycoside (digitalis, digoxin), statin, antipsychotic (neuroleptic), tricyclic antidepressant, selective serotonin reuptake inhibitor, other antidepressant, benzodiazepine, opioid, antiepileptic. Assessed through the electronic health record
Fall-risk increasing drugs | Day 30 (+/-5) after enrollment
  Including loop diuretic, beta blocker, cardiac glycoside (digitalis, digoxin), statin, antipsychotic (neuroleptic), tricyclic antidepressant, selective serotonin reuptake inhibitor, other antidepressant, benzodiazepine, opioid, antiepileptic. Assessed by telephone interview of the participant
Fall-risk increasing drugs | Day 180 (+/-5) after enrollment
  Including loop diuretic, beta blocker, cardiac glycoside (digitalis, digoxin), statin, antipsychotic (neuroleptic), tricyclic antidepressant, selective serotonin reuptake inhibitor, other antidepressant, benzodiazepine, opioid, antiepileptic. Assessed by telephone interview of the participant
Number of patients with fall(s) during hospitalization (hospitalization duration expected to be 3 to 20 days on average) | Discharge (-1 to +2 days after discharge)
  Based on nurse report and electronic health record data
Number of falls per patient during hospitalization (hospitalization duration expected to be 3 to 20 days on average) | Discharge (-1 to +2 days after discharge)
  Based on nurse report and electronic health record data
Number of patients with fall(s) within 30 days after discharge | Day 30 (+/-5) after enrollment
  Assessed by telephone interview of the participant/relatives, based on a diary the participants/relatives will be asked to complete.
Number of falls per patient within 30 days after discharge | Day 30 (+/-5) after enrollment
  Assessed by telephone interview of the participant/relatives, based on a diary the participants/relatives will be asked to complete.
Number of patients with fall(s) within 180 days after discharge | Day 180 (+/-5) after enrollment
  Assessed by telephone interview of the participant/relatives, based on a diary the participants/relatives will be asked to complete.
Number of falls per patient within 180 days after discharge | Day 180 (+/-5) after enrollment
  Assessed by telephone interview of the participant/relatives, based on a diary the participants/relatives will be asked to complete.
Number of patients with new institutionalization at discharge | Discharge (-1 to +2 days after discharge)
  According to nurses / electronic health record / self-report by participant/relatives
Number of patients with new institutionalization within 30 days of discharge | Day 30 (+/-5) after enrollment
  Assessed by telephone interview of the participant/relatives
Number of patients with new institutionalization within 180 days of discharge | Day 180 (+/-5) after enrollment
  Assessed by telephone interview of the participant/relatives
Number of patients with emergency room visits within 30 days of discharge | Day 30 (+/-5) after enrollment
  Assessed based on electronic health record and by telephone interview of the participant/relatives, based on the diary the participant/relatives will be asked to complete.
Number of emergency room visits per patient within 30 days of discharge | Day 30 (+/-5) after enrollment
  Assessed based on electronic health record and by telephone interview of the participant/relatives, based on the diary the participant/relatives will be asked to complete.
Number of patients with emergency room visits within 180 days of discharge | Day 180 (+/-5) after enrollment
  Assessed based on electronic health record and by telephone interview of the participant/relatives, based on the diary the participant/relatives will be asked to complete.
Number of emergency room visits per patient within 180 days of discharge | Day 180 (+/-5) after enrollment
  Assessed based on electronic health record and by telephone interview of the participant/relatives, based on the diary the participant/relatives will be asked to complete.
Number of patients with readmission within 30 days of discharge | Day 30 (+/-5) after enrollment
  Assessed based on electronic health record and by telephone interview of the participant/relatives, based on the diary the participant/relatives will be asked to complete.
Number of readmissions per patient within 30 days of discharge | Day 30 (+/-5) after enrollment
  Assessed based on electronic health record and by telephone interview of the participant/relatives, based on the diary the participant/relatives will be asked to complete.
Number of patients with readmission within 180 days of discharge | Day 180 (+/-5) after enrollment
  Assessed based on electronic health record and by telephone interview of the participant/relatives, based on the diary the participant/relatives will be asked to complete.
Number of readmissions per patient within 180 days of discharge | Day 180 (+/-5) after enrollment
  Assessed based on electronic health record and by telephone interview of the participant/relatives, based on the diary the participant/relatives will be asked to complete.
Experience of the intervention | Discharge (-1 to +2 days after discharge)
  Assessed through qualitative and quantitative questions by interview of the participants/relatives (on the ward or by telephone). For the intervention group only. Will be done at the end of the assessment to preserve outcome assessor blinding.
Satisfaction with hospitalization | Discharge (-1 to +2 days after discharge)
  Measured by the satisfaction questionnaire adapted and simplified
Perspectives on hospital mobility | Day 30 (+/-5) after enrollment
  Quantitative questions (Likert-scale answers) based on the Health Action Process Approach (HAPA) model (simplification of a survey used in the preparation phase of this study to assess perspectives of patients and healthcare professionals on hospital mobility).
Location at follow-up | Day 30 (+/-5) after enrollment
  Assessed by telephone interview of patient/relatives.
Location at follow-up | Day 180 (+/-5) after enrollment
  Assessed by telephone interview of patient/relatives.
Discharge destination | Discharge (-1 to +2 days after discharge)
  Assessed based on electronic health records

OTHER OUTCOMES:
Healthcare professional experience of the intervention and perspectives on hospital mobility | After cluster closure (on average 1 to 10 months, maximum 15 months)
  Semi-structured interview and survey (in the intervention group only)
Patient opinion on comfort and practicability of the StepWatch and GENEActiv accelerometers | Discharge (-1 to +2 days after discharge)
  Outcome of the pilot study only. Assessment through semi-structured interview
Patient opinion on comfort and practicability of the ActiGraph accelerometer | Discharge (-1 to +2 days after discharge)
  Outcome of the randomized trial only. Assessment through semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Carole E Aubert, MD, MSc, Principal Investigator — Bern University Hospital, Inselspital, University of Bern, Bern, Switzerland
Locations (4):
- Switzerland (4):
  - Kantonsspital Baden, Baden, Canton of Aargau
  - HFR-Fribourg - hôpital cantonal, Villars-sur-Glâne, Canton of Fribourg
  - Spital Tiefenau, InselGruppe AG, Bern
  - Inselspital, Bern University Hospital, InselGruppe AG, Bern

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan, informed consent form will be published. Other data will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After study completion
Access Criteria: Upon reasonable request

REFERENCES:
- [Derived] Mooser B, Bergsma D, Liechti FD, Baumgartner C, Gentizon J, Mean M, Wertli MM, Mancinetti M, Schmidt-Leuenberger J, Aubert CE. Impact of an INtervention to increase MOBility in older hospitalized medical patients (INTOMOB): Study protocol for a cluster randomized controlled trial. BMC Geriatr. 2023 Oct 31;23(1):705. doi: 10.1186/s12877-023-04285-3. PMID 37907858

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT05639231/SAP_000.pdf